CLINICAL TRIAL: NCT01916863
Title: A Phase 1, Single-center, Partially Double-blind, Randomized, Single-dose, 3-Period Crossover Study to Assess the Pharmacodynamic Effects of LX4211 and INVOKANA™ (Canagliflozin) in Healthy Subjects Using Stable Isotope Tracer Methods
Brief Title: Study to Evaluate the Effect of Single Doses of LX4211 and Canagliflozin on Intestinal Glucose Absorption in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LX4211.1-111-NRM; LX4211.111 (Other: Lexicon Pharmaceuticals, Inc.)
Record Dates: First submitted 2013-07-29; First posted 2013-08-06 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol; Canagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- LX4211 (Experimental): 400 mg of LX4211
  Interventions: Drug: LX4211 400 mg; Drug: canagliflozin 300 mg; Drug: LX4211 Placebo
- Canagliflozin (Active Comparator): 300 mg canagliflozin
  Interventions: Drug: LX4211 400 mg; Drug: canagliflozin 300 mg; Drug: LX4211 Placebo
- Placebo (Placebo Comparator): LX4211 placebo
  Interventions: Drug: LX4211 400 mg; Drug: canagliflozin 300 mg; Drug: LX4211 Placebo

INTERVENTIONS:
Drug: LX4211 400 mg
Drug: canagliflozin 300 mg
Drug: LX4211 Placebo

SUMMARY:
The purpose of this study is to assess the effect of LX4211 and the comparator drug canagliflozin on intestinal glucose absorption and metabolism after a single dose in healthy subjects in comparison to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects ≥18 to ≤55 years of age
* Vital signs at Screening in the following ranges: systolic blood pressure, 90-140 mmHg; diastolic blood pressure, 50-90 mmHg; heart rate, 45-100 bpm
* Body mass index (BMI) ≥18 and ≤35 kg/sq m
* Willing and able to provide written informed consent

Exclusion Criteria:

* Use of any medication (prescription, over-the-counter, herbal tea, or supplements) within 7 days of dosing
* Use of any investigational agent or study treatment within 30 days of Day -1
* Use of any protein or antibody-based therapeutic agents within 3 months of Screening
* Prior exposure to LX4211 or canagliflozin
* Daily use of >5 cigarettes or any tobacco products within 6 weeks prior to Screening and while participating in the study
* History of bariatric surgery or any other gastrointestinal surgery that may induce malabsorption
* History of bowel resection, any malabsorptive disorder, severe gastroparesis, any GI procedure for the purpose of weight loss which would slow gastric emptying
* History of any major surgery within 6 months prior to Screening
* History of any hypersensitivity to the inactive components of LX4211, inactive components of canagliflozin, acetaminophen oral solution or any inactive component of acetaminophen liquid preparation
* History of renal disease or significantly abnormal kidney function tests
* History of hepatic disease or significantly abnormal liver function tests
* History of any active infection within 30 days prior to Day -1
* History of alcohol or substance abuse within 2 years prior to Day 1
* History of hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab), HIV-1 or HIV-2
* Donation or loss of >500 mL of blood or blood product within 56 days of Day -1
* positive pregnancy test at Screening or Day -1
* Positive urine screen for drugs of abuse at Screening or Day -1
* Positive breath test for alcohol at Screening or Day -1
* Inability or difficulty swallowing whole tablets
* Unable or unwilling to communicate or cooperate with the Investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2013-08; Primary Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in rate of glucose appearance after meal (RaO) | Days 1, 8, 15

SECONDARY OUTCOMES:
Rate of total glucose appearance (RaT) | Days 1, 8, 15
Change from baseline in fasting plasma glucose | Days 1, 8, 15
Change from baseline in postprandial glucose | Days 1, 8, 15
Change from baseline in insulin | Days 1, 8, 15

CONTACTS AND LOCATIONS:
Overall Officials: Paul Strumph, M.D., Study Director — Lexicon Pharmaceuticals, Inc.
Locations (1):
- Lexicon Investigational Site, Chula Vista, California, United States

REFERENCES:
- [Derived] Powell DR, Zambrowicz B, Morrow L, Beysen C, Hompesch M, Turner S, Hellerstein M, Banks P, Strumph P, Lapuerta P. Sotagliflozin Decreases Postprandial Glucose and Insulin Concentrations by Delaying Intestinal Glucose Absorption. J Clin Endocrinol Metab. 2020 Apr 1;105(4):e1235-49. doi: 10.1210/clinem/dgz258. PMID 31837264